CLINICAL TRIAL: NCT02715193
Title: A Randomized, Placebo-controlled, Double-blind, In-patient Study to Evaluate Safety, Tolerability, and Pharmacodynamics of REMD-477 Following a Single Dose in Subjects With Type 1 Diabetes Mellitus
Brief Title: Single-dose Study to Evaluate Safety, Tolerability, and Pharmacodynamics of REMD-477 in Subjects With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: REMD Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R477-101
Record Dates: First submitted 2016-02-29; First posted 2016-03-22 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Type 1 Diabetes Mellitus; Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — volagidemab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- REMD-477 Treatment A (Experimental): Administered as a single SC dose in subjects with Type 1 Diabetes
  Interventions: Biological: REMD-477
- Matching placebo (Placebo Comparator): Administered as a single SC dose in subjects with Type 1 Diabetes
  Interventions: Biological: Placebo Comparator

INTERVENTIONS:
Biological: REMD-477
  Arms: REMD-477 Treatment A
Biological: Placebo Comparator
  Arms: Matching placebo

SUMMARY:
This is a randomized, placebo-controlled, double-blind study to evaluate safety, tolerability and pharmacodynamics of REMD-477 in subjects who have Type 1 diabetes and are currently receiving insulin treatment. This proof of concept study will determine whether glucagon receptor blockade using a single dose REMD-477 can improve short-term glucose homeostasis in people with Type 1 diabetes.

DETAILED DESCRIPTION:
The study will be conducted at two sites in the United States, and approximately 20 subjects with type 1 diabetes will be enrolled. Eligible subjects will be admitted to the clinical research unit, to carefully monitor blood glucose; and establish the baseline insulin requirement for maintaining targeted normoglycemia (postabsorptive: 90-120 mg/dL; and postprandial: <180 mg/dL).

The patients will then be subjected to a hyperglycemic period (250-300 mg/dL) by a stepwise reduction in insulin infusion. After receiving a single SC dose of REMD-477 or matching placebo in a double-blinded fashion, all subjects will be assessed for the post-treatment 24-hour insulin requirement needed to maintain targeted normoglycemia (postabsorptive: 90-120 mg/dL; and postprandial: <180 mg/dL); and to be monitored closely for safety, tolerability and targeted glycemic control, for a 48-hr period. After the in-patient residency period, subjects will return to the clinic for weekly out-patient safety follow-up visits for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 18 and 60 years old, inclusive, at the time of screening;
* Females of non-child bearing potential must be ≥1 year post-menopausal (confirmed by a serum follicle-stimulating hormone (FSH) levels ≥ 40 IU/mL) or documented as being surgically sterile. Females of child bearing potential must agree to use two methods of contraception;
* Male subjects must be willing to use clinically acceptable method of contraception during the entire study;
* Body mass index between 18.5 and 26.9 kg/m2, inclusive, at screening;
* Diagnosed with Type 1 diabetes for greater than 2 years, based on clinical history or as defined by the current American Diabetes Association (ADA) criteria;
* HbA1c ≥6.0 % but <9.0 % at screening;
* Fasting C-peptide <0.2 ng/mL;
* Current use of insulin pump and willing to use continuous glucose monitoring (CGM) system (e.g. DexCom) throughout the entire study;
* ALT and/or AST within <1.5x ULN at screening;
* Serum amylase and lipase within normal limits at screening;
* Able to provide written informed consent approved by an Institutional Review Board (IRB).

Exclusion Criteria:

* History or evidence of clinically-significant disorder or condition that, in the opinion of the Investigator, would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion;
* Significant organ system dysfunction (e.g., clinically significant pulmonary or cardiovascular disease, anemia [Hemoglobin <10.0 g/dL], and renal dysfunction [eGFR <90 ml/1.73M2/min]);
* Any severe symptomatic hypoglycemic event associated with a seizure or requiring help from other people or medical facility in the past 6 months;
* Current or recent (within 1 month of screening) use of diabetes medications other than insulin;
* Use of steroids and/or other prescribed or over-the-counter medications that are known to affect the outcome measures in this study or known to influence glucose metabolism;
* Smokes tobacco;
* Known sensitivity to mammalian-derived drug preparations, recombinant protein-based drugs or to humanized or human antibodies;
* History of illegal drug use or alcohol abuse within the last 6 months or a positive drug urine test result at screening;
* History of pancreatitis, pancreatic neuroendocrine tumors or multiple endocrine neoplasia;
* History of pheochromocytoma, or family history of familial pheochromocytoma;
* Known or suspected susceptibility to infectious disease (eg, taking immunosuppressive agents or has a documented inherited or acquired immunodeficiency);
* Positive for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HbsAg), or hepatitis C antibodies (HepC Ab);
* Participation in an investigational drug or device trial within 30 days of screening or within 5 times the half-life of the investigational agent in the other clinical study, if known, whichever period is longer;
* Blood donor or blood loss >500 mL within 30 days of Day 1;
* Women who are pregnant or lactating/breastfeeding;
* Regular exercise >120 min/week within 14 days of Day 1;
* Unable or unwilling to follow the study protocol or who are non-compliant with screening appointments or study visits;
* Family history of multiple endocrine neoplasia.

Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events per subject, including changes in vital signs, physical and neurological examinations, laboratory safety tests and ECGs | Baseline and 57 days
Changes from baseline in 24-hour insulin requirements on Day 1 relative to the two 24 hour periods post-treatment on Days 3 and 4, between the REMD-477 and placebo treated subjects, needed to maintain targeted glycemic control. | Baseline (24 hour period on Day 1) and Days 3 and 4

SECONDARY OUTCOMES:
Immunogenicity: Incidence of REMD-477 neutralizing and non-neutralizing antibodies | Baseline and 57 days
Changes from baseline over time of AST. | Baseline and 57 days
  Incidence of elevated serum aspartate transaminase (AST) values > 3x the upper limit of normal (ULN).
Changes from baseline over time of ALT. | Baseline and 57 days
  Incidence of elevated serum alanine transaminase (ALT) values >3x the upper limit of normal (ULN).
Changes from baseline over time of ALP. | Baseline and 57 days
  Incidence of elevated serum alkaline phosphatase (ALP) >2x upper limit of normal (ULN)
Changes from baseline over time of total bilirubin. | Baseline and 57 days
  Incidence of elevated serum total bilirubin >2x upper limit of normal (ULN).
Changes from baseline over time of amylase | Baseline and 57 days
  Incidence of elevated serum amylase values at >2.5x ULN
Changes from baseline over time of lipase | Baseline and 57 days
  Incidence of elevated serum lipase values at >2.5x ULN

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - San Diego, California
  - St Louis, Missouri

REFERENCES:
- [Derived] Pettus J, Reeds D, Cavaiola TS, Boeder S, Levin M, Tobin G, Cava E, Thai D, Shi J, Yan H, Bautista E, McMillan J, Unger R, Henry RR, Klein S. Effect of a glucagon receptor antibody (REMD-477) in type 1 diabetes: A randomized controlled trial. Diabetes Obes Metab. 2018 May;20(5):1302-1305. doi: 10.1111/dom.13202. Epub 2018 Jan 22. PMID 29283470